CLINICAL TRIAL: NCT04547335
Title: The Influence of CYP2C19 Polymorphisms on the Safety and Efficacy of Voriconazole in Adult Patients With Hematologic Malignancy Receiving Voriconazole Treatment Due to an Invasive Fungal Infection
Brief Title: The Influence of CYP2C19 Polymorphisms on the Safety and Efficacy of Voriconazole
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Principal Investigator, Mukaddes Gumustekin, Full Professor, Dokuz Eylul University
Other Study IDs: 19-AKD-47
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Adverse Drug Reactions
Keywords: voriconazole; invasive aspergillosis; adverse drug reactions; CYP2C19 polymorphisms; pharmacogenetics; hematologic malignancy; efficacy
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Hematologic Neoplasms | interventions — Voriconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 9 mL of blood sample collected into an EDTA (Ethylenediaminetetraacetic Acid) tube for PGx analysis
  9 mL of blood sample collected into an EDTA (Ethylenediaminetetraacetic Acid) tube for voriconazole TDM
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Voriconazole: All eligible patients will be followed up for voriconazole related adverse drug events and efficacy
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — This is an observational study and only the patients already on voriconazole treatment will be included in the study.

SUMMARY:
Voriconazole is a drug used to treat invasive fungal infections. The amount of voriconazole in a person's blood helps to determine how effectively it treats an infection, and how safe it is. Patients respond differently when receiving the same dose - some clearly benefit, other patients experience side effects, and others see limited improvement in their infection.

Voriconazole is broken down in the liver mainly by an enzyme called CYP2C19, before being excreted from the body. The activity of CYP2C19 differs between people because of variation in the DNA that encodes the body's instructions to make CYP2C19.

If CYP2C19 activity is very high, voriconazole blood levels may remain below the target range when a patient receives a standard dose of voriconazole, which may be insufficient to treat their infection. By contrast, decreased CYP2C19 activity due to genetic variation may result in excessively high voriconazole blood levels, predisposing to serious side effects.

Therefore, knowing a patient's CYP2C19 genetic makeup is very important for predicting their response to voriconazole. Thus, the investigators aim to determine the influence of genetic variation in CYP2C19 on the frequency and severity of side effects related to voriconazole, and on the effectiveness of voriconazole for treating serious fungal infections. The findings from this study will contribute to determining the optimal dose of voriconazole that patients with different genetic variants in CYP2C19 should be started on, and will take us one step closer to both understanding the genetic structure of CYP2C19 in the Turkish population, and to 'personalised medicine'.

DETAILED DESCRIPTION:
Rationale for the study:

Although the incidence of invasive aspergillosis (IA) in patients with hematological malignancies has decreased by half, its mortality rate still remains of substantial clinical concern.

Voriconazole is the first line therapy for the treatment of IA. Since it has a narrow therapeutic window, the high inter/intra-individual variability and nonlinear pharmacokinetics, therapeutic drug monitoring (TDM) is recommended to optimize clinical outcomes. Voriconazole is metabolized principally by CYP2C19 (cytochrome P450 enzyme) and, to a lesser extent, by CYP3A4 and CYP2C9 enzymes. Among the various covariates, CYP2C19 genetic variability is the major determinant that contributes to interindividual variability of voriconazole. While the poor metabolizers are more susceptible to toxicity, the risk of treatment failure in ultra-metabolizers are considered to be higher. TDM improve the safety and efficacy of voriconazole treatment. The appropriate time for TDM is after the first few days (2-5 days) of initiation of standard treatment. However some adverse drug reactions (ADRs) and deviation from the therapeutic range may occur until the TDM is done. Starting with pharmacogenetic-guided dose would ensure safer and more effective therapy until the TDM is performed and would lead to less frequent TDM with decreased treatment costs. Furthermore, pharmacogenetic test results can also be used when interpreting the optimal dose of other drugs that is metabolized with the same enzyme. The individual pharmacogenetic data also enables safer and cost-effective therapy adjustments in the future, too.

Therefore, primary objective of the study is to determine the influence of CYP2C19 genetic polymorphisms on the frequency and severity of ADRs related to voriconazole during the study period in a Turkish university hospital. The secondary objective is to determine the influence of CYP2C19 genetic polymorphisms on the effectiveness of voriconazole in this setting. Our study will fill this gap by assessing the influence of CYP2C19 polymorphisms on the safety and efficacy of voriconazole that is being used in patients with a hematologic malignancy to treat an IA.

1.Methods

The study population will be drawn from patients aged 18 and over that are hospitalized in Dokuz Eylul University Hospital Hematology Service due to a hematological malignancy, and are receiving voriconazole for the management of an IFI, which is diagnosed based on EORTC/MSG ( European Organisation for Research and Treatment of Cancer / Mycosis Study Group) criteria.

1.1.Data and sample collection

1.1.1.Data collection: At baseline, demographics and clinical information will be recorded from all patients directly and complemented from their medical records. All patients will be followed up by the research team daily for the first 7 days following voriconazole initiation, and then on days 14, 30 and 60. All follow up will be initially via assessment of medical records, with additional data input from the patient directly. The medical records include: the electronic hospital record system (PROBEL), paper-based patient records and other patient follow-up- documents.

During routine clinical care, ADRs are monitored daily by a hematology fellow and/or an infectious disease specialist. On days one to seven following voriconazole initiation, the investigators will record these clinical evaluations daily; they will also capture these data on days 14 and 30.

For participants that had either started voriconazole active treatment before they were recruited, or were recruited during the maintenance phase of their voriconazole regimen, the research team will assess their medicals records retrospectively between the point of recruitment and day one of their active voriconazole treatment to detect ADRs.

On days 30 and 60, patient survival will be recorded by review of patient records only.

Treatment response (efficacy) will be determined based on the EORTC/MSG consensus criteria 30. These data will be obtained at all follow up points (from day one to seven, and days 14, 30 and 60).

The follow-up scheme and the consort flow diagram regarding the protocol are attached in the appendix.

1.1.2.Sample collection: 1.1.2.1.Samples fo PGx analysis: For PGx analysis, participants will donate one 9 mL blood sample collected into an EDTA (Ethylenediaminetetraacetic Acid) tube on day one whilst blood samples are being taken from the patient for daily routine clinical purposes (without requiring any other needle insertion). Samples for PGx analysis will be coded and stored securely in the Department of Medical Pharmacology at the DEUTF. The samples will be stored -80 celsius degree until used up. PGx analysis will be performed in the Department of Molecular and Clinical Pharmacology at the University of Liverpool at the end of the study. Participants and physicians will not be informed of the participant's genotype as this is an observational study. The participant's clinical care will not be affected in any way by taking part in the study

1.1.2.2.Samples for voriconazole concentration determination The second 9 mL blood sample will be collected into a red cap tube on the fifth day (9th dose) of treatment before the morning voriconazole dose, again whilst blood is being collected as part of routine clinical care (without requiring any other needle insertion) to determine the trough voriconazole concentration at steady state. This blood sample will be centrifuged and the serum stored in the Department of Medical Pharmacology at the Dokuz Eylul University Faculty of Medicine. When follow up is completed for a given patient, this serum sample will be transferred to an accredited laboratory in Istanbul, Turkey, with maintenance and assurance of the cold chain during sample transportation to guarantee sample integrity.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Receiving voriconazole for the treatment of an invasive fungal infection (IFI) and are within the first five days of the treatment course, OR are receiving voriconazole for the secondary prophylaxis against IFI during or after chemotherapy
* Agree to give one additional blood sample twice during the study for the purposes of pharmacogenetic analysis and determination of the serum trough voriconazole concentration, whilst their blood is being collected during normal clinical follow up without the requirement for any additional intravenous intervention
* Are willing and able to give informed consent and sign the informed consent form

Exclusion Criteria:

* Have previously had CYP2C19 PGx testing performed
* Pregnant/breastfeeding
* Have cognitive impairment and/or psychiatric disorders and/or any other condition that will draw into question their capacity to provide informed consent
* Have severe hepatic insufficiency (Child-Pugh Class C) and have renal failure (estimated GFR <15ml/min /1,73m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 and over that are hospitalized in Dokuz Eylul University Hospital Hematology Service due to a hematological malignancy, and are receiving voriconazole for the management of IFI, which is diagnosed based on EORTC/MSG criteria
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of voriconazole related adverse drug reactions | Follow up period for primary outcome is 30 days for each participant
  Voriconazole related adverse drug reactions of grade 3-5 systematically evaluated using Liverpool Causality Assessment Tool identified during study follow up.
  Severity of all adverse events will be graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0

SECONDARY OUTCOMES:
Non-response to voriconazole | Follow up period for this outcome is 60 days for each participant
  The efficacy of voriconazole treatment will be assessed based on reviews of clinical, mycological and radiological data according to the Mycoses Study Group and European Organization for Research and Treatment of Cancer Consensus Criteria (EORTC/MSG criteria).
Voriconazole trough concentration | 30 minutes before the 9th dose of voriconazole
  Voriconazole trough concentration will be measured once for each participant from plasma samples collected 30 minutes before the 9th dose of voriconazole
Survival | On days 30 and 60
  Patient survival will be evaluated on days 30 and 60 by reference to the Dokuz Eylul University Hospital Hematology Service; date of death will be captured to permit survival analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mukaddes Gumustekin, Professor, MD, PhD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided